CLINICAL TRIAL: NCT03043846
Title: Treat to Target Trial in Axial Spondylo Arthritis : The TICOSPA (Tight Control in Spondyloarthritis)
Acronym: TICOSPA
Status: Completed | Type: Observational
Sponsor: Association de Recherche Clinique en Rhumatologie (Other)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-A00564-47
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Axial Spondyloarthritis
Keywords: Treat to Target approach
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tight control and Treat to Target arm: For this group, the treating rheumatologist will agree to monitor very closely (at least every 4 weeks) and also to treat their patients in accordance with a pre-defined strategy.
  Interventions: Other: Follow-up every 3 months during 1 year (data collection in eCRF); Other: Follow-up every month to follow the pre-defined strategy
- Usual care arm: For this arm, the treating rheumatologists will continue to manage the enrolled patients in accordance to their usual care.
  Interventions: Other: Follow-up every 3 months during 1 year (data collection in eCRF)

INTERVENTIONS:
Other: Follow-up every 3 months during 1 year (data collection in eCRF)
Other: Follow-up every month to follow the pre-defined strategy
  Groups: Tight control and Treat to Target arm

SUMMARY:
This is a not interventional, pragmatic, prospective, randomized (cluster) study to evaluate the potential benefit of a Treat to Target approach in comparison to routine treatment (i.e. usual care) in patients with axial spondyloarthritis.

DETAILED DESCRIPTION:
This study is reflecting the usual care either in accordance to the treating rheumatologist (arm: usual care) or in accordance to the international scientific recommendations (arm: T2T)

The tight control means that as soon as a treatment is initiated in a patient, the time permitting to evaluate its potential efficacy/safety has to be determined. In terms of safety, such time frame can be very short based on the occurrence of adverse events. In terms of efficacy it is usually recommended to evaluate an NSAIDs after 2 to 4 weeks of treatment intake and the TNF blockers after 12 to 16 weeks.

The Treat to Target means that there is an a priori decision of the target to reach while initiating a treatment and more importantly an a priori decision to intensify the treatment in case such target is not achieved.

There will be 2 arms in the study (tight control and treat to target arm and usual care arm).

160 patients (80 patients per arm) will be included during one year by 18 centers (10 in France, 4 in Belgium and 4 in Netherlands). Patients will be followed during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adults (between 18 and 65 years old)
* With a diagnosis of axial spondyloarthritis according to the axial ASAS criteria AND the opinion of the treating rheumatologist.
* Active disease defined as an ASDAS ≥ 2.1
* Predominant axial disease meaning that:

  * Patients with non-spinal rheumatological symptoms and/or extra-rheumatological manifestations requiring at baseline the initiation of a specific treatment will be excluded.
  * Patients with a past history and/or a current well controlled non-spinal rheumatological or extra-rheumatological features will be eligible for the study.
* Non-optimally treated with NSAIDs (i.e. who have not received at least 2 NSAIDS, daily during at least 2 weeks at full dose, during the last year). Annex II summarizes the list of commonly used NSAIDs and the definition of a "full" use.
* With available pelvic X-rays, B27 and MRI of the sacro-iliac joints (performed at any time since symptoms onset)
* With no contraindication to the use of a NSAID
* With no intake of apremilast during the previous 3 months
* Able to understand the objectives of the study and to fill the questionnaires
* Written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosis of predominant axial spondyloarthritis according to the axial ASAS criteria AND the opinion of the treating rheumatologist, and an active disease defined as an (ASDAS ≥ 2.1), and non-optimally treated with NSAIDs.
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
To compare the changes in ASASHI-NRS over the one year of follow-up in the 2 groups | After a one year follow-up
  In the original protocol, the main objective was "to compare the percentage of patients with a significant improvement in the ASAS-HI score after a one year follow-up in the 2 groups".
  However, after further research on the methodology to better assess the treatment effect on a pragmatic cluster-based strategy trial, we propose to change the primary objective for two reasons in order to:
  * Calculate a "significant improvement" of the ASAS-HI, we would need to be aware of the minimally clinically important difference, and this threshold has not been yet defined for the regular ASAS-HI nor for the ASAS-HI NRS.
  * Account for the reduced heterogeneity induced by the fact that patients are clustered, a multilevel analysis (e.g. mixed models with two random effects, the subject and the cluster or center) has been proposed as the most appropriate method.
  Therefore, we have amended the main objective to: "To compare the changes in ASASHI-NRS over the one year of follow-up in the 2 groups".

SECONDARY OUTCOMES:
To compare the percentage of patients reaching an ASDAS major improvement after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the percentage of patients reaching an ASDAS clinically important improvement after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the percentage of patients reaching a BASDAI 50 after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the change in the ASDAS over one year follow-up in the 2 groups. | After a one year follow-up
To compare the change in the BASDAI over one year follow-up in the 2 groups. | After a one year follow-up
To compare the change in the ASAS-NSAID score over one year follow-up in the 2 groups. | After a one year follow-up
To compare the WPAI after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the EQ5D after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the self-report questionnaire on health resource utilization after a one year follow-up in the 2 groups. | After a one year follow-up
To compare the number and type of adverse events occuring over one year follow-up in the 2 groups. | After a one year follow-up
To compare the treatment effect (...) within the T2T depending on the compliance to the T2T treatment. | After a one year follow-up

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (4):
  - UZ GENT, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Reumatologie Medizorg, Merksem
  - AZ Alma, Sijsele
- France (10):
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - Chu Le Mans, Le Mans
  - Hopital Lapeyronnie, Montpellier
  - Ch Mulhouse, Mulhouse
  - Hopital Cochin, Paris
  - Hopital de La Pitie Salpetriere, Paris
  - Hopital Henri Mondor, Paris
  - Chu Rouen, Rouen
  - Chu Toulouse, Toulouse
- Netherlands (4):
  - UMCG, Groningen
  - Zuyderland MC, Heerlen
  - LUMC, Leiden
  - Maastricht UMC, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molto A, Lopez-Medina C, Van den Bosch FE, Boonen A, Webers C, Dernis E, van Gaalen FA, Soubrier M, Claudepierre P, Baillet A, Starmans-Kool M, Spoorenberg A, Jacques P, Carron P, Joos R, Lenaerts J, Gossec L, Pouplin S, Ruyssen-Witrand A, Sparsa L, van Tubergen A, van der Heijde D, Dougados M. Efficacy of a tight-control and treat-to-target strategy in axial spondyloarthritis: results of the open-label, pragmatic, cluster-randomised TICOSPA trial. Ann Rheum Dis. 2021 Nov;80(11):1436-1444. doi: 10.1136/annrheumdis-2020-219585. Epub 2021 May 6. PMID 33958325